CLINICAL TRIAL: NCT06848205
Title: Basal Ganglia Contributions to Transitions in Freezing of Gait and Parkinson's Disease
Brief Title: Percept Transitions in FOG and PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NEUR-2024-33357; STUDY00023279 (Other: University of Minnesota)
Record Dates: First submitted 2025-02-19; First posted 2025-02-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Freezing of Gait; Parkinson Disease
Keywords: FOG; PD; Freezing of Gait; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: In the second experiment: we will compare LFPs during the successful movement transitions vs. freezing-events during a FOG provocation course in people with FOG only.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's disease with freezing of gait (Experimental): Participants will have a Medtronic Percept DBS device, diagnosis of idiopathic Parkinson's disease (PD), and freezing of gait (FOG).
  Interventions: Other: OFF Parkinson's Medication(s); Other: OFF Deep Brain Stimulation
- Parkinson's disease without freezing of gait (Experimental): Participants will have a Medtronic Percept DBS device and diagnosis of idiopathic Parkinson's disease (PD) without having freezing of gait (FOG).
  Participants in this arm will not be tested in experiment #2.
  Interventions: Other: OFF Parkinson's Medication(s); Other: OFF Deep Brain Stimulation

INTERVENTIONS:
Other: OFF Parkinson's Medication(s) — Participants will be asked to withhold Parkinson's medications 12 hours prior to their testing visit (if extended-release Parkinson's medications are taken by the participant, they will be asked to withhold these for 24 hours prior to their testing visit).
Other: OFF Deep Brain Stimulation — Participants will have their deep brain stimulation turned off at the beginning of their testing visit.

SUMMARY:
The purpose of this research is to examine the possible causes and signs of freezing of gait (FOG) secondary to Parkinson's disease (PD). To achieve this, the study will use the novel (on-label and FDA-approved) local field potential (LFP) measuring capability of the Medtronic Percept™ deep brain stimulation (DBS) system to compare oscillatory activity in people who have Parkinson's disease, with and without freezing of gait (FOG). This will be conducted as three separate experiments, participants may volunteer for one or more experiments:

Experiment 1: The first experiment will compare LFPs during gait initiation with and without a cue, in people with (PD+FOG) and without FOG (PD-FOG).

Experiment 2: The second experiment will compare LFPs during the successful movement transitions vs. freezing-events during a FOG provocation course in people with FOG.

Experiment 3: The third experiment will compare LFPs during rapid alternating movements of the wrist and/or foot, in people with and without FOG

DETAILED DESCRIPTION:
The purpose of this research is to examine the underlying pathophysiology and biomarkers of freezing of gait (FOG) and cueing-evoked improvements. This protocol will use the novel (on-label, FDA-approved) local field potential (LFP)-measuring capability of the Medtronic Percept™ deep brain stimulation (DBS) system to compare oscillatory activity in people who have Parkinson's disease (PD), with and without freezing of gait (FOG). This will be conducted as three separate experiments, participants may volunteer for one or more experiments:

Experiment 1: The first experiment will compare LFPs during gait initiation with and without a cue, in people with (PD+FOG) and without FOG (PD-FOG).

Experiment 2: In the second experiment, the investigators will compare LFPs during the successful movement transitions vs. freezing-events during a FOG provocation course in people with FOG.

Experiment 3: In the third experiment, the investigators will compare LFPs during rapid alternating movements of the wrist and/or foot, in people with and without FOG.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD.
* Age 21-75 (see Inclusion of Individuals across the Lifespan for justification of age range).
* Able to ambulate independently without the use of an assistive device (e.g. cane) for 50 meters.
* Implanted Medtronic Percept TM Device.
* At least 3 months since the initial activation of the neurostimulator.
* Undervalued, under-represented, or disenfranchised social group may be included.
* Active members of the military (service members), DoD personnel (including civilian employees) may be included.
* Individual or group that is disadvantaged in the distribution of social goods and services such as income, housing, or healthcare may be included.

Exclusion Criteria:

* Meet criteria for dementia with Lewy bodies, Multiple Systems Atrophy, Alzheimer's disease, or other neurodegenerative disorder.
* History of seizures or other significant neurological disorders that may affect participation or performance in the study.
* History of musculoskeletal disorders that significantly affect walking or movement of limb(s) that would affect the participation in the experimental task (Participants will be excluded from that task, but may participate in other tasks, for example, may be excluded from Experiment 1 if the disorder affects walking, but may still participate in Experiment 3).
* History of muscular conditions of the neck and back, including whiplash that would affect walking experiments.
* History of visual and/or vestibular conditions that may affect participation or performance in the study.
* Reduced capacity to consent. This will be assessed using a 2-stage process. Initially, participants will be tested using the University of California, San Diego, Brief Assessment of Capacity to Consent (UBACC). If concerns are raised from the UBACC test, the individual will be further tested using the MacArthur Competency Assessment Tool.
* Pregnant people.
* Post-operative complications or adverse effects (e.g. ON stimulation dystonia) that affect patient safety or confound the experiment.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of the anticipatory postural adjustments magnitudes (cm) | During the intervention
  Blocks of 10 successful step initiation trials will be performed. Ground reaction forces (Kistler Inc.) will be recorded.
Quantification of the anticipatory postural adjustments duration (sec) | During the intervention
  Blocks of 10 successful step initiation trials will be performed. Ground reaction forces (Kistler Inc.) will be recorded.
Step characteristics of the first two steps, length (cm) | During the intervention
  Blocks of 10 successful step initiation trials will be performed. Ground reaction forces (Kistler Inc.) and bipolar surface electromyographic (EMG) signals will be recorded bilaterally from seven muscles (tibialis anterior, soleus, lateral gastrocnemius, rectus femoris, biceps femoris, semimembranosus, gluteus medius) (Delsys, Trigno) at 1000 Hz and synchronized to whole body kinematics (8-camera motion capture system, SIMI Inc. or Qualisys Inc.) collected at 100 or 120 Hz and with 128-channels of EEG data (BioSemi, Amsterdam) collected at 2000 Hz according to the 10:20 international system 35. Additionally, resting-state EEG will be collected, to reference and remove walking artifact 36 . Local field potentials (LFPs) will be recorded on the Medtronic Percept system and synchronized to the other data collection systems by briefly turning the device on and off.
Step characteristics of the first two steps, width (cm) | During the intervention
  Blocks of 10 successful step initiation trials will be performed. Ground reaction forces (Kistler Inc.) and bipolar surface electromyographic (EMG) signals will be recorded bilaterally from seven muscles (tibialis anterior, soleus, lateral gastrocnemius, rectus femoris, biceps femoris, semimembranosus, gluteus medius) (Delsys, Trigno) at 1000 Hz and synchronized to whole body kinematics (8-camera motion capture system, SIMI Inc. or Qualisys Inc.) collected at 100 or 120 Hz and with 128-channels of EEG data (BioSemi, Amsterdam) collected at 2000 Hz according to the 10:20 international system 35 . Additionally, resting-state EEG will be collected, to reference and remove walking artifact 36 . Local field potentials (LFPs) will be recorded on the Medtronic Percept system and synchronized to the other data collection systems by briefly turning the device on and off.
Step characteristics of the first two steps, duration (sec) | During the intervention
  Blocks of 10 successful step initiation trials will be performed. Ground reaction forces (Kistler Inc.) and bipolar surface electromyographic (EMG) signals will be recorded bilaterally from seven muscles (tibialis anterior, soleus, lateral gastrocnemius, rectus femoris, biceps femoris, semimembranosus, gluteus medius) (Delsys, Trigno) at 1000 Hz and synchronized to whole body kinematics (8-camera motion capture system, SIMI Inc. or Qualisys Inc.) collected at 100 or 120 Hz and with 128-channels of EEG data (BioSemi, Amsterdam) collected at 2000 Hz according to the 10:20 international system 35 . Additionally, resting-state EEG will be collected, to reference and remove walking artifact 36 . Local field potentials (LFPs) will be recorded on the Medtronic Percept system and synchronized to the other data collection systems by briefly turning the device on and off.
The coherence magnitudes between the cortex and globus pallidus (dB) | During the intervention
  Blocks of 10 successful step initiation trials will be performed. Ground reaction forces (Kistler Inc.) and bipolar surface electromyographic (EMG) signals will be recorded bilaterally from seven muscles (tibialis anterior, soleus, lateral gastrocnemius, rectus femoris, biceps femoris, semimembranosus, gluteus medius) (Delsys, Trigno) at 1000 Hz and synchronized to whole body kinematics (8-camera motion capture system, SIMI Inc. or Qualisys Inc.) and with 128-channels of EEG data (BioSemi, Amsterdam) collected at 2000 Hz according to the 10:20 international system 35. Additionally, resting-state EEG will be collected, to reference and remove walking artifact 36. Local field potentials (LFPs) will be recorded on the Medtronic Percept system and synchronized to the other data collection systems by briefly turning the device on and off. Coherence will be calculated between the cortex and basal ganglia, and the magnitudes will be calculated at different frequencies (power, decibels, dB).
The coherence magnitudes between the cortex and EMG (dB) | During the intervention
  Blocks of 10 successful step initiation trials will be performed. Ground reaction forces (Kistler Inc.) and bipolar surface electromyographic (EMG) signals will be recorded bilaterally from seven muscles (tibialis anterior, soleus, lateral gastrocnemius, rectus femoris, biceps femoris, semimembranosus, gluteus medius) (Delsys, Trigno) at 1000 Hz and synchronized to whole body kinematics (8-camera motion capture system, SIMI Inc. or Qualisys Inc.) and with 128-channels of EEG data (BioSemi, Amsterdam) according to the 10:20 international system 35 . Additionally, resting-state EEG will be collected, to reference and remove walking artifact 36 . Local field potentials (LFPs) will be recorded on the Medtronic Percept system and synchronized to the other data collection systems by briefly turning the device on and off. Coherence will be calculated between the cortex and the muscle activity, and the magnitudes will be calculated at different frequencies (power, decibels, dB).
The coherence magnitudes between the globus pallidus and EMG (dB) | During the intervention
  Blocks of 10 successful step initiation trials will be performed. Ground reaction forces (Kistler Inc.) and bipolar surface electromyographic (EMG) signals will be recorded bilaterally from seven muscles (tibialis anterior, soleus, lateral gastrocnemius, rectus femoris, biceps femoris, semimembranosus, gluteus medius) (Delsys, Trigno) at 1000 Hz and synchronized to whole body kinematics (8-camera motion capture system, SIMI Inc. or Qualisys Inc.) and with 128-channels of EEG data (BioSemi, Amsterdam) according to the 10:20 international system 35 . Additionally, resting-state EEG will be collected, to reference and remove walking artifact 36 . Localfield potentials (LFPs) will be recorded on the Medtronic Percept system and synchronized to the other data collection systems by briefly turning the device on and off. Coherence will be calculated between the globus pallidus and the muscle activity, and the magnitudes will be calculated at different frequencies (power, decibels, dB).
Number of freezing episodes | During the intervention
  Kinematics will be measured using 6 inertial measurement units (IMUs, Opal sensors, APDM), containing triaxial accelerometers, gyro-scopes, and magnetometers, on each foot and wrist, the fifth lumbar vertebra, and the sternum. This system has been validated for use in PD gait to provide measures of gait (velocity, stride length mean and SD, cadence, and stride time mean and SD), gait initiation (measures of APA and 1 st step characteristics) and turning. Kinematic data will be collected at 128 Hz and synchronized to video recordings and LFP data. LFP and kinematic data will be classified by transition type: initiation, turning, and doorways, and compared during successful transitions, and freezing episodes (unsuccessful transitions). Number of freezing episodes will be identified and rated qualitatively from the videotape by a blinded rater.
Rapid Alternating Movements of Wrist Pronation/Supination (degrees) | During the intervention
  Participants will perform rapid alternating movements of the wrist or ankle while a manipulandum measures their angular position, with EMG of the moving limb, EEG and LFPs are recorded synchronously. Movements will be cued using a series of beeps that will change randomly between a low and a high- frequency. RMS of the amplitude will be calculated.
Rapid Alternating Movements of Supination or Ankle plantar/dorsi-flexion (degrees) | During the intervention
  Participants will perform rapid alternating movements of the wrist or ankle while a manipulandum measures their angular position, with EMG of the moving limb, EEG and LFPs are recorded synchronously. Movements will be cued using a series of beeps that will change randomly between a low and a high- frequency. RMS of the amplitude will be calculated.
Peak power of local field potential oscillations (dB) | During the intervention
  Average changes in peak alpha and beta power derived from power spectral density analysis of the local field potential signal recorded by the implanted Medtronic Percept™ device.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Movement Disorders Lab, Minneapolis, Minnesota, United States